CLINICAL TRIAL: NCT07169812
Title: Investigation of the Relationship Between Vertical Jump, Balance, Muscle Strength, Flexibility, and Foot Posture in Artistic Gymnasts
Brief Title: Relationship Between Vertical Jump, Balance, Muscle Strength, Flexibility, and Foot Posture in Artistic Gymnasts
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Gülenay Yıldırım, PhD Student, Istanbul University - Cerrahpasa
Other Study IDs: ICU2025-06
Record Dates: First submitted 2025-09-03; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Vertical Jump; Dynamic Balance; Flexibility; Foot Posture Index Score; Muscle Strength
Keywords: dynamic balance; flexibility; foot posture index; muscle strength; vertical jump

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Artistic gymnastics is a highly demanding and technically complex sport that requires strength, flexibility, agility, balance, and coordination (Nassib et al., 2020). Gymnasts perform a series of dynamic movements, such as flips, turns, and somersaults, which require explosive muscular power and precise control (Potop et al., 2014). In this sport, jumping ability, balance, muscle strength, and flexibility are fundamental physical parameters that directly influence both movement quality and injury risk. Among these, jumping ability plays a particularly critical role by facilitating take-offs and aerial maneuvers, enabling gymnasts to generate the necessary height and momentum to perform complex routines effectively. Moreover, gymnasts with greater jump capacity are able to absorb landings more efficiently, thereby reducing injury risk and maintaining consistent performance throughout their routines (Feng et al., 2024; Geiblinger et al., 2025).

Another essential parameter is balance-particularly dynamic balance, which can be defined as the body's ability to perceive and respond to postural changes that occur during motor activities. This involves maintaining the center of mass within the base of support, requiring a high level of neuromuscular activation. Dynamic balance is vital not only in sports but also in daily life activities such as walking, stair climbing, running, and sit-to-stand transitions. Its role in preventing injuries and enhancing athletic performance has been well established (Paillard, 2019; Dana et al., 2021). The Y-Balance Test (YBT), which measures dynamic balance in three directions-anterior (ANT), posterolateral (PL), and posteromedial (PM)-is commonly used in clinical and athletic settings. In clinical practice, a difference of less than 4 cm between limbs in each direction is considered normative. Lehr et al. (2013) reported in a study conducted among collegiate athletes that average YBT performance could serve as a predictor of future lower extremity injuries.

From a biomechanical perspective, the foot represents the distal segment of the lower extremity kinetic chain. Any morphological changes or alterations in the weight-bearing alignment of the foot can influence balance control. Considering the critical role of the foot in stabilizing and modulating the kinetic chain, accurately assessing foot posture is essential. Postural characteristics such as high or low arches may impact balance capacity, jump performance, and the ability to attenuate forces during landing (Seyedahmadi et al., 2024).

In light of this evidence, the primary aim of the present study is to examine the relationships between vertical jump performance, balance, muscle strength, flexibility, and foot posture in artistic gymnasts. Investigating these parameters comprehensively is expected to provide valuable insights from both scientific and clinical perspectives.

Specifically, the study seeks to: Determine the relationship between vertical jump performance and lower extremity muscle strength, flexibility, and balance. Analyze the potential associations between foot posture and vertical jump, balance, and muscle strength. By addressing these objectives, the study aims to contribute to both guiding the design of training programs and reducing the risk of injury among gymnasts, thereby offering meaningful clinical implications.

This is an observational, cross-sectional study. Participants will continue their regular gymnastics training routines without any intervention assigned by the investigators. Data collection will consist solely of measurements (vertical jump, balance, muscle strength, flexibility, and foot posture). No exercise program, treatment, or intervention will be applied as part of the study.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study. Participants will continue their regular gymnastics training routines without any intervention assigned by the investigators. Data collection will consist solely of measurements (vertical jump, balance, muscle strength, flexibility, and foot posture). No exercise program, treatment, or intervention will be applied as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in artistic gymnastics for 1-2 years
* Age between 7 and 12 years

Exclusion Criteria:

* History of lower extremity orthopedic injury within the past 6 months
* Presence of any pain at the time of assessment
* History of neurological, developmental, or systemic disease that may affect balance
* Uncorrectable visual impairments
* Obesity or any neurological or musculoskeletal abnormality that could affect postural stability
* Voluntary withdrawal from the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will include healthy child athletes aged 7-12 years who have been actively participating in artistic gymnastics training for 1-2 years at gymnastics clubs.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump | Baseline
  The active vertical jump performance of participants will be evaluated using the My Jump Lab (MJL) mobile application. My Jump Lab is a practical and portable tool with established validity and reliability. In a validity-reliability study conducted by Balsalobre-Fernández et al. (2024), Cronbach's α was reported to be greater than 0.93. Similarly, Şentürk et al. (2024) compared the application with a force platform and demonstrated an almost perfect correlation between the two methods (r = 0.968, p = 0.001), confirming that MJL is a valid and reliable instrument for real-time assessment of jump performance and active jump height.
  Each participant will complete three practice trials at their perceived maximum effort prior to testing. The MJL application will be used on an iPhone 14 (Apple Inc., Cupertino, CA, USA). To record active jump height, the iPhone will be mounted on a tripod positioned to capture the participant's sagittal plane. Participants will be instructed to place their h

SECONDARY OUTCOMES:
Dynamic Balance | Baseline
  Dynamic balance of the participants will be evaluated using the Y-Balance Test (YBT), which is a modified version of the Star Excursion Balance Test. The YBT has been shown to be valid and reliable, with intrarater ICC values ranging from 0.85 to 0.91 and interrater ICC values between 0.99 and 1.00 (Plisky et al., 2009). The test can be performed on the floor or with a custom apparatus, consisting of a Y-shaped system extending in three directions: anterior, posteromedial, and posterolateral. The posteromedial and posterolateral arms are positioned at a 90° angle relative to each other, and both form 135° angles with the anterior arm.
  During the test, children will stand at the center of the Y with their hands on their hips, balancing on the dominant leg while reaching in the anterior, posteromedial, and posterolateral directions with the opposite leg, touching the furthest possible point with their toe while maintaining balance. Each direction will be tested three times for both limb
Muscle Strength | Baseline
  Isolated muscle strength will be assessed using the Lafayette Model 01165A Manual Muscle Testing System, a portable digital hand-held dynamometer with an LCD display and three interchangeable heads (Instrument, 2012). The device provides measures such as peak force, time to peak force, total test duration, and average force in kilograms, Newtons, or pounds.
  Measurements will be performed by the same investigator, using the same hand, three times for both dominant and non-dominant lower limbs. The mean value will be used as the final muscle strength score. Maximum isometric strength of bilateral the hip flexors, extensors, abductors and adductors as well as the knee flexors and extensors, will be measured using the "make" test protocol with the digital dynamometer.
Foot Posture | Baseline
  Foot posture will be assessed using the Foot Posture Index-6 (FPI-6), developed by Redmond et al. (2006). The FPI-6 evaluates foot posture based on six criteria: palpation of the talar head, observation of supra- and infra-malleolar curvature, calcaneal frontal plane position, prominence of the navicular region, congruence of the medial longitudinal arch, and forefoot abduction/adduction. Each item is scored from -2 (indicating supination) to +2 (indicating pronation), with the total score indicating overall foot posture.
  Scores from 0 to +5 represent neutral alignment, positive values above +5 indicate pronation, and negative values below 0 indicate supination. The Turkish version of the FPI-6 has demonstrated excellent reliability, with internal consistency coefficients of Cronbach's α = 0.85 and 0.78, test-retest reliability ICC(2,k) = 0.96 and 0.94, and inter-rater reliability ICC(2,k) = 0.93 for both dominant and non-dominant lower extremities (Yağcıoğlu et al., 2024).

OTHER OUTCOMES:
Flexibility | Baseline
  Flexibility in the sagittal plane will be evaluated using the Sit-and-Reach Test. Participants will be seated with their feet flat against a fixed surface, ankles in a neutral position, and knees fully extended. They will be instructed to reach forward with their hands, keeping their knees extended, and touch as far as possible. The distance reached by the third finger will be measured with a tape measure. Scores beyond the toes will be recorded as positive values, while scores short of the toes will be recorded as negative. The test will be repeated three times, and the best score will be recorded in centimeters (Castro-Piñero et al., 2009).

IPD SHARING:
Plan to Share IPD: No